CLINICAL TRIAL: NCT04673916
Title: Analysis of the Efficacy of Two Treatment Protocols for Patients With Symptomatic Oral Lichen Planus
Brief Title: Treatment Protocols for Patients With Symptomatic Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121/120/PO
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Lichen Planus, Oral; Preneoplastic Condition
MeSH Terms: conditions — Lichen Planus, Oral; Precancerous Conditions

STUDY DESIGN:
Intervention Model Description: 2 groups of patients
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clobetasol treatment (Active Comparator): The clobetasol group was treated with clobetasol propionate 0.05%, while the anti-inflammatory group was treated with mouthwash. The drug used consisted of Clobetasol propionate 0.05%, Ethyl alcohol 96° (50%), Hydroxyethylcellulose (4%); Preserved water (just enough to 100%) that was topically applied [11]. This drug was produced as a galenic formulation. Clobetasol propionate twice a day (every 12 hours) to the lesions with a soft bristle brush and were advised not to drink or eat during the hour following application of the medication.
  Interventions: Drug: Healing evaluation
- Anti-inflammatory mouthwash (Active Comparator): In patients of the anti-inflammatory group, the mouthwash was used pure and without dilution at a dosage of 20 ml 3 times a day, immediately after normal daily oral hygiene was prescribed. It contains calcium hydroxide, hyaluronic acid, Umbelliferone and Oligomeric Proanthocyanidins. Patients were instructed to rinse for at least 5 minutes over the entire oral mucosa, with particular emphasis on the regions where the lesions are located.
  Interventions: Drug: Healing evaluation

INTERVENTIONS:
Drug: Healing evaluation — Treatments were topically applied for 5 days

SUMMARY:
The primary objective of this study was to compare the therapeutic efficacy of clobetasol propionate 0.05% oral gel versus an anti-inflammatory mouthwash in an oral solution for the management of patients suffering from symptomatic OLP. The secondary objective was to analyze which one of the two treatments induced a greater risk of developing side effects.

DETAILED DESCRIPTION:
Forty patients were assigned (20 patients per group), through a randomized design, to receive clobetasol (clobetasol gel 0.05%), or an anti-inflammatory mouthwash (mouthwash which contains calcium hydroxide, hyaluronic acid, Umbelliferone and Oligomeric Proanthocyanidins) for 3-months. At baseline (T0) and after 3 months (T1), patients were subjected to clinical and oral assessments and were evaluated for the symptoms (Numerical Pain Scale, NRS score) and signs (Thongprasom's score) of OLP. Data were calculated using T-test for the dependent variable, Wilcoxon test and Mann-Witney u test.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* clinical diagnosis and histological diagnosis of OLP on the basis of WHO criteria;
* presence of symptoms related to OLP.

Exclusion Criteria:

* presence of systemic conditions that may have affected the study results;
* state of pregnancy or breastfeeding;
* histological signs of dysplasia;
* drugs inducing a lichen response (ACE-inhibitors, β-blockers, etc.);
* treatment of OLP in the six months prior to the start of the programme;
* presence of extraoral lesions (genital, skin and other)
* history of previous immunodeficiency or HIV seropositivity;
* previous allogeneic bone marrow transplantation;
* presence of systemic lupus erythematosus or other autoimmune diseases.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Clinical Mucosal healing | 180 days
  Patients clinically were evaluated using the scale used by Thongprasom et al. as reference. This gives a score that varies from 0 to 5, using a millimetre reference: 0, in the absence of lesions; 1, in the presence of hyperkeratosis streaks; 2, in the presence of an atrophic area less than 1 mm2; 3, in the presence of an atrophic area greater than 1 mm2; 4, in the presence of an erosive area less than 1 mm2; 5, in the presence of an erosive area greater than 1 mm2. In the presence of multiple injuries, the value has been calculated by summing the values of each injury.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing clinical results
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: University website and pubmed

REFERENCES:
- [Derived] Santonocito S, Polizzi A, De Pasquale R, Ronsivalle V, Lo Giudice A, Isola G. Analysis of the Efficacy of Two Treatment Protocols for Patients with Symptomatic Oral Lichen Planus: A Randomized Clinical Trial. Int J Environ Res Public Health. 2020 Dec 23;18(1):56. doi: 10.3390/ijerph18010056. PMID 33374791